CLINICAL TRIAL: NCT03480412
Title: Repeated Luteal Phase Ovarian Stimulation (Second Step Protocol) in Poor Responder Patients
Brief Title: Second Step Protocol in Poor Ovarian Responder (POR)
Acronym: POR
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Università degli Studi 'G. d'Annunzio' Chieti e Pescara (Other)
Responsible Party: Principal Investigator, Antonia Iacovelli, Doctor, Università degli Studi 'G. d'Annunzio' Chieti e Pescara
Other Study IDs: Second Step 1
Record Dates: First submitted 2018-03-21; First posted 2018-03-29 (Actual); Last update posted 2018-04-02 (Actual); Status verified 2018-03

CONDITIONS: Infertility, Female; Premature Ovarian Failure; Fertility Disorders
Keywords: Luteal Phase Stimulation; Poor Ovarian Response; In Vitro Fertilization
MeSH Terms: conditions — Infertility, Female; Primary Ovarian Insufficiency | interventions — Follicular Phase; Luteal Phase

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Follicular Phase
  Interventions: Procedure: Follicular Phase
- Luteal Phase
  Interventions: Procedure: Luteal Phase

INTERVENTIONS:
Procedure: Follicular Phase — The follicular phase stimulation is conduced according to a standardized Antagonist protocol or Short protocol (with GnRH agonist) using recombinant or urinary gonadotropins (starting dose 300 or 450 UI) or a long lasting recombinant gonadotropin (Corifollitropin alfa 150 mcg) from the second day of the menstrual cycle. When at least two follicles had reached 17-18 mm in diameter, ovulation will be triggered with a single subcutaneous bolus of urinary human chorionic gonadotropin (10.000 UI ) and oocyte retrieval will be performed after 35 hours.
  Other Names: First Step
  Groups: Follicular Phase
Procedure: Luteal Phase — Two - six days after the first oocyte retrieval a second gonadotropin stimulation will be started with a GnRH antagonist protocol (the stimulation will be started with 250 UI of human menopausal gonadotropin (hMG) and a GnRH antagonist (GnRH-an) 0,25 mg\die will be administered when the leading follicle is ≥ 14 mm until hCG criteria are met). When at least two follicles had reached 17-18 mm in diameter, ovulation will be triggered with a single subcutaneous bolus of urinary human chorionic gonadotropin (10.000 UI ) and oocyte retrieval will be performed after 35 hours.
  Other Names: Second Step
  Groups: Luteal Phase

SUMMARY:
Reduced ovarian reserve and the consequent poor ovarian response are very recurent in infertile patients, indeed a percentage of 10%-24% of couples addressed to infertility program may be classified as Poor Ovarian Responder (POR).

Objective: To evaluate whether the repeated luteal phase stimulation (Second Step) permits a significantly higher number of oocytes retrieved in POR when compared to conventional follicular stimulation.

Interventions: The follicular phase stimulation is conduced according to a standardized Antagonist protocol or Short protocol (with GnRH agonist) using recombinant or urinary gonadotropins (starting dose 300 or 450 UI) or a long lasting recombinant gonadotropin (Corifollitropin alfa 150 mcg).

Two - six days after the first oocyte retrieval a second gonadotropin stimulation will be started with a GnRH antagonist protocol (the stimulation will be started with 250 UI of human menopausal gonadotropin (hMG) and a GnRH antagonist (GnRH-an) 0,25 mg\die will be administered when the leading follicle is ≥ 14 mm until hCG (human chorionic gonadotropin) criteria are met. When at least two follicles had reached 17-18 mm in diameter, ovulation will be triggered with a single subcutaneous bolus of urinary human chorionic gonadotropin (10.000 UI ) and oocyte retrieval will be performed after 35 hours.

Two or Three months after the second oocyte retrieval the Embryo transfer (ET) will be performed after endometrial preparation with Estradiol Valerate and intramuscular Progesterone.

DETAILED DESCRIPTION:
Reduced ovarian reserve and the consequent poor ovarian response are very recurent in infertile patients, indeed a percentage of 10%-24% of couples addressed to infertility program may be classified as Poor Ovarian Responder (POR).

Poor ovarian response and reduced ovarian reserve can be caused by different factors such as advanced female age, smoking, autoimmune diseases, aneuploidies and genetic diseases or can be idiopathic.

An Eshre ( European Society of Human Reproduction and Embryology) consensus in 2011 established the "Bologna Criteria" that consented a standardize definition of poor ovarian response (POR).

According with the Bologna Criteria we can diagnose a Poor Ovarian Response or an expected Poor Ovarian Response when at least two of the following three features are present:

* Advanced maternal age (≥40 years) or any other risk factor for POR;
* A previous POR (≤3 oocytes with a conventional stimulation protocol);
* An abnormal ovarian reserve test (i.e. AFC -Antral Follicular Count- 5-7 follicles or AMH ,0.5-1.1 ng/ml). The diagnosis and the prediction of poor ovarian response consent the selection of the best treatment with the aim of the retrieval of an high number of oocytes.

A lot of treatment have been proposed to optimize in vitro fertilization outcomes in POR (high dosage of Gonadotropins; short protocol, administration of androgens or Aromatase Inhibitors, administration of Growth Hormone and the repeated luteal phase stimulation).

The Luteal Phase Stimulation was initially proposed for fertility preservation procedures, but in last years is used in POR patients too. The recently diffused "wave theory" support this technique. According to the wave theory two or three cohorts of antral follicles are recruited during the follicular and luteal phase of each ovarian cycle and in one of this follicular wave will be selected the dominant follicle.

A trial performed in 2014 (Kuang et al, 2014) pubblished results of repeated luteal phase stimulation (Shanghai Protocol) showing that double ovarian stimulations in the same menstrual cycle provide more opportunities for retrieving oocytes in poor responders. More recently another trial (Ubaldi et al 2016) did not observe significant differences in term of number of oocytes retrieved and euploid blastocyst rate from follicular versus luteal phase stimulation.

Objective: To evaluate whether the repeated luteal phase stimulation (Second Step) permits a significantly higher number of oocytes retrieved in POR when compared to conventional follicular stimulation.

Interventions: The follicular phase stimulation is conduced according to a standardized Antagonist protocol or Short protocol (with GnRH agonist) using recombinant or urinary gonadotropins (starting dose 300 or 450 UI) or a long lasting recombinant gonadotropin (Corifollitropin alfa 150 mcg) from the second day of the menstrual cycle. When at least two follicles had reached 17-18 mm in diameter, ovulation will be triggered with a single subcutaneous bolus of urinary human chorionic gonadotropin (10.000 UI ) and oocyte retrieval will be performed after 35 hours.

Two - six days after the first oocyte retrieval a second gonadotropin stimulation will be started with a GnRH antagonist protocol (the stimulation will be started with 250 UI of human menopausal gonadotropin (hMG) and a GnRH antagonist (GnRH-an) 0,25 mg\die will be administered when the leading follicle is ≥ 14 mm until hCG criteria are met). When at least two follicles had reached 17-18 mm in diameter, ovulation will be triggered with a single subcutaneous bolus of urinary human chorionic gonadotropin (10.000 UI ) and oocyte retrieval will be performed after 35 hours.

Two or Three months after the second oocyte retrieval the Embryo transfer (ET) will be performed after endometrial preparation with Estradiol Valerate and intramuscular Progesterone.

ELIGIBILITY:
Inclusion Criteria:

* Antral Follicular Count ≤7 follicles
* Number of oocyte retrieved with First oocyte retrieval ≤ 2

Exclusion Criteria:

* Antral follicular Count < 7
* Anti-Müllerian hormone (AMH) >1.1 ng \mL
* Number of oocyte retrieved with First oocyte retrieval > 2
* Absence of antral follicles after First oocyte retrieval

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Women classified like Poor Ovarian Responder
Study Population: Infertil Women classified as Poor Ovarian Responder according with Bologna Criteria (2011) for which an IVF is indicated and in which the number of oocyte retrieved with First oocyte retrieval ≤ 2
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2017-09-01 (Actual); Primary Completion 2019-03-30 (Estimated); Study Completion 2019-09 (Estimated)

PRIMARY OUTCOMES:
Number of oocyte Retrieved | 15 days after the Second oocyte retrieval
  Number of oocyte Retrieved after the first oocyte retrieval vs Number of oocyte Retrieved after the second oocyte retrieval

SECONDARY OUTCOMES:
Number of Embryos Obtained | 15 days after the Second oocyte retrieval
  Number of Embryos Obtained after the Follicular Phase Stimulation and intracytoplasmic sperm injection vs Number of Embryos obtained after Luteal Phase Stimulation and intracytoplasmic sperm injection

CONTACTS AND LOCATIONS:
Locations (1):
- Ospedale G. Bernabeo, Ortona, Chieti, Italy